CLINICAL TRIAL: NCT01961375
Title: MIRENA for Contraception In InDian Subjects User continuAtion and Satisfaction Study.
Brief Title: MIRENA for Contraception In InDian Subjects User continuAtion and Satisfaction Study: MIDAS Study
Acronym: MIDAS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16199; MA1210IN (Other: company internal)
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: BAY 86-5028; Levonorgestrel- Intra Uterine System
  Interventions: Drug: Levonorgestrel- Intra Uterine System (BAY 86-5028_Mirena)

INTERVENTIONS:
Drug: Levonorgestrel- Intra Uterine System (BAY 86-5028_Mirena) — Levonorgestrel 52 mg intrauterine system with release rate of upto 20 mcg/day, Intrauterine insertion

SUMMARY:
The study is designed as non interventional to observe the continuation rate and the patient satisfaction in women who have a LNG-IUS (Levonorgestrel releasing Intrauterine system) inserted for contraception over the period of 12 months under real life condition in India.The study will begin after the study approval by ethics committee.All Indian women aged between 18-49 years who are initiating LNG IUS therapy for contraception will be included in study after taking the informed consent.Patients will be observed for upto 12 months.The study involves general examination of patients, collection of data like medical history, previous contraceptive use,concomitant medication etc.The study is planned to enroll 600 subjects from multiple study centers spread across India. The study data will be analyzed with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 18-49 years who are initiating LNG IUS therapy for contraception.
* Subject willing to provide informed consent and comply with study procedure.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study subjects will be enrolled from multiple sites like women's hospitals, tertiary care institutes, Family planning clinics and gynaecological consulting centres.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Percentage continuation rate of LNG IUS at end of observation period. | 12 months
Percentage of Women with user satisfaction scoring somewhat satisfied to very satisfied | 12 months

SECONDARY OUTCOMES:
Cumulative discontinuation rate for pregnancy | 12 months
Cumulative discontinuation rate for other medical reasons | 12 months
Cumulative discontinuation rate for non-medical reasons | 12 months
Mean percentage of women with amenorrhea | 12 months
Mean percent of women with spotting, inter-menstrual bleeding | 12 months
Distribution of contraceptive usage patterns | 12 months
  contraceptive usage patterns included:birth-spacing, long term contraception, postpartum contraception, post-abortion contraception, switch from other method, contraception for other medical reasons like heart disease, etc
Incidence rate of drug-related adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.